CLINICAL TRIAL: NCT05042453
Title: Prospective, Multicenter, 60 Months, Single-arm Cohort Trial for Evaluation of the Efficacy and Safety of Transvaginal Sacrospinous Ligament Fixation With Splentis for the Treatment of Primary Apical Pelvic Organ Prolapse
Brief Title: Long-term Evaluation of the Efficacy and Safety of Splentis for the Treatment of Primary Apical Pelvic Organ Prolapse
Acronym: SAXO
Status: Recruiting | Type: Observational
Sponsor: Promedon (Industry)
Responsible Party: Sponsor
Other Study IDs: Sax_Pro
Record Dates: First submitted 2021-08-12; First posted 2021-09-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Apical Pelvic Organ Prolapse; Transvaginal repair; Mesh augmented repair; Sacrouterine ligament fixation
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hysteropexy using Splentis via vaginal route: Non-fertile women ≥ 18 years with uterine descent (POP-Q ≥ 2) which are study-independently scheduled for hysteropexy with Splentis
  Interventions: Device: Splentis® POP Tissue Anchoring System

INTERVENTIONS:
Device: Splentis® POP Tissue Anchoring System — Anterior cervicopexy with bilateral sacrospinous ligament fixation using Splentis

SUMMARY:
This prospective, multi center cohort trial aims to evaluate the efficacy and safety of hysteropexy using Splentis via the vaginal route in primary uterine prolapse

DETAILED DESCRIPTION:
Women who undergo hysteropexy with Splentis via the vaginal route for primary uterine prolapse will be evaluated regarding efficacy and safety in a long term follow-up of 60 months. The primary endpoint is composed of anatomical, subjective and re-treatment components, whereas several secondary endpoints focusing on functional outcome including overactive bladder symptoms, urinary incontinence, quality of life and sexual life will be considered. Furthermore, a detailed report about adverse events will be included.

ELIGIBILITY:
Inclusion Criteria:

* non-fertile women
* primary symptomatic uterine descent POP-Q≥2
* Scheduled apical POP repair with Splentis
* Willing and able to participate at study visits and to sign informed consent

Exclusion Criteria:

* Fertile women
* Recurrent apical prolapse
* Women with post hysterectomy vaginal vault prolapse
* Patients with active or latent infection of the vagina, cervix or uterus
* Patients with previous or current vaginal, cervical or uterine cancer
* Previous, current or planned pelvic radiation therapy
* Known allergy to polypropylene.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-fertile women ≥ 18 years with uterine prolapse
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Cure of apical pelvic organ prolapse | 12 months
  Cure of apical pelvic organ prolapse is defined according the current recommendations by Barber et al. and ICS/IUGA recommendations. Therefore, a combined endpoint using anatomical, subjective and necessity retreatment criteria are utilized.
  Primary endpoint is the number of patients achieving all criteria of the composite endpoint:
  1. leading edge of the apical vaginal wall at or above the hymen (C≤ 0)
  2. absence of a vaginal bulge symptom
  3. no need for retreatment of the apical prolapse by either pessary use or surgical intervention

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, 6 weeks 12, 24, 36, 60 months
  Change of Quality of life and prolapse symptoms using the Prolapse-Quality of Life-Questionnaire in comparison between baseline and follow-up.
  The questionnaire is divided in nine domains which are analyzed separately. The results will be transformed into a scale between 0 - 100 according the questionnaires description. The higher the score, the higher the impact of prolapse symptoms and the lower the quality of life.
Quality of life | Baseline, 6 weeks and 12, 24, 36, 60 months
  Change of quality of life using the EQ-5L-5D in comparison between baseline and follow-up.
  It consists of a 5-item descriptive system as well as a visual analogue scale ranging from 0 to 100. It is conceptualized to assess deviation from health and hereby provide health related quality of life problems.
Urinary incontinence | Baseline, 6 weeks and 12, 24, 36, 60 months
  Change of urinary incontinence using the International Consultation on Incontinence Questionnaire- Urinary Incontinence Short From in comparison between baseline and follow-up
  The ICIQ-UI-SF includes four items with a sum score ranging between 0 and 21 points. The higher the score the higher the impact of symptoms.
Overactive Bladder | Baseline, 6 weeks and 12, 24, 36, 60 months
  Change of urinary incontinence using the International Consultation on Incontinence Questionnaire- Overactive bladder in comparison between baseline and follow-up
  The score of the ICIQ-OAB ranges from 0 to 16 points. The higher the sum score the higher the impact of symptoms.
Sexual life | Baseline, 6 weeks and 12, 24, 36, 60 months
  Change of sexual life using the Pelvic Organ Prolapse Incontinence Sexual Questionnaire- IUGA revised in comparison between baseline and follow-up.
  The result will be transformed into a scale between 0 - 100. The higher the score, the higher the impact of prolapse symptoms and the higher the impact on sexual life.
Pain according Visual analogue scale of pain | Baseline, 24-48 hours postoperatively, 6 weeks and 12, 24, 36, 60 months
  Change of pain using the visual analogue scale of pain in comparison between baseline and follow-up
  The Wong-Baker Faces Pain Scale is a visual analogue scale to assess subject pain.The answers will be transformed in a scale from 0 to 10 whereas 0 implicate no pain and 10 worst pain.
Patient global impression of improvement | 6 weeks and 12, 24, 36, 60 months
  Number of Patients with improvement of prolapse symptoms according the validated question Patient Global Impression of improvement
  The PGI-I is a seven Likert scale from very much better to no change and very much worse.
Cure according composite endpoint | 6 weeks and 24, 36, 60 months
  Number of patients completing each component of the composite endpoint
Adverse Events | Intraoperatively, 24-48hours postoperatively, 6 weeks postoperatively and 12, 24, 36, 60 months, unscheduled visits
  Number and severity of Adverse Events according guideline of AE reporting, Clavien Dindo and Terminology of IUGA/ICS
Exposure and extrusion free survival | 6 weeks and 12, 24, 36, 60 months
  Estimated exposure and extrusion free survival according Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Naumann, MD, Principal Investigator — Helios Clinic Erfurt, Germany; Christian Fünfgeld, MD, Principal Investigator — Clinic Tettnang
Locations (7):
- Germany (7):
  - DRK Hospital Chemnitz-Rabenstein, Chemnitz
  - Helios Hospital Erfurt, Department of gynaecology, Erfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - Clinic Kassel, Kassel
  - St. Elisabeth Hospital, Leipzig
  - University Hospital, Mannheim
  - Hospital Tettnang, Tettnang

IPD SHARING:
Plan to Share IPD: No